CLINICAL TRIAL: NCT05573568
Title: Inhaled N, N-Dimethyltryptamine: a Phase I Study in Healthy Adults
Brief Title: Clinical Study of DMT in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biomind Labs Inc. (Industry)
Collaborators: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BMND01
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
Keywords: N,N-DMT; DMT; N,N-Dimethyltryptamine; Healthy Volunteers
MeSH Terms: interventions — N,N-Dimethyltryptamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A - single ascending dose (Experimental): Administration of up to 2 inhaled doses of DMT within a single day (5 mg, followed by 20 mg) with a 2-hour dose interval (5 subjects).
  Interventions: Drug: N,N-Dimethyltryptamine
- Group B - single ascending dose (Experimental): Administration of up to 2 inhaled doses of DMT within a single day (7.5 mg, followed by 30 mg) with a 2-hour dose interval (5 subjects).
  Interventions: Drug: N,N-Dimethyltryptamine
- Group C - single ascending dose (Experimental): Administration of up to 2 inhaled doses of DMT within a single day (10 mg, followed by 40 mg) with a 2-hour dose interval (5 subjects).
  Interventions: Drug: N,N-Dimethyltryptamine
- Group D - single ascending dose (Experimental): Administration of up to 2 inhaled doses of DMT within a single day (12.5 mg, followed by 50 mg) with a 2-hour dose interval (5 subjects).
  Interventions: Drug: N,N-Dimethyltryptamine
- Group E - single ascending dose (Experimental): Administration of up to 2 inhaled doses of DMT within a single day (15 mg, followed by 60 mg) with a 2-hour dose interval (5 subjects).
  Interventions: Drug: N,N-Dimethyltryptamine

INTERVENTIONS:
Drug: N,N-Dimethyltryptamine — DMT will be administered using a vaporizer device in a single ascending fixed-order dosing regimen
  Other Names: DMT; BMND01

SUMMARY:
This study aims to evaluate the acute and subacute effects of an inhaled N, N-Dimethyltryptamine in healthy individuals.

DETAILED DESCRIPTION:
Participants will receive N, N-Dimethyltryptamine administered in two dosing sessions: an initial low-dose safety session and subsequent intermediate-dose treatment, in a fixed order and 2h apart.

ELIGIBILITY:
Inclusion Criteria:

* prior experience with N,N-Dimethyltryptamine (DMT)
* present proof of vaccination against COVID-19 (Coronavírus)

Exclusion Criteria:

* heart failure
* liver failure
* kidney failure
* resistant hypertension
* arrhythmia
* valvular heart disease
* chronic obstructive pulmonary disease
* asthma
* severe obesity
* epilepsy
* pregnancy
* thyroid disorders
* family diagnosis or suspicion of genetic monoamine oxidase deficiency
* previous adverse response to psychedelic substances
* present or past symptoms or family members with a psychotic disorder
* dissociative identity disorder
* bipolar disorder
* prodromal symptoms of schizophrenia
* abuse of alcohol or other psychoactive substances, except tobacco
* acute or sub-acute risk of suicide
* flu-like symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as clinical and psychiatry symptoms assessed by qualitative medical/clinical-psychiatry evaluation | up to 1 month after dosing
  Evaluate clinical and psychiatry acute risks after DMT treatments assessed by qualitative medical evaluation after dosing.
Blood Pressure | up to 2 hours after each dose
  Assessed 20 times on each dose via systolic and diastolic blood pressure
Heart rate | up to 2 hours after each dose
  Assessed 20 times on each dose
Respiratory rate | up to 2 hours after each dose
  Assessed 20 times on each dose
Oxygen saturation | up to 2 hours after each dose
  Assessed 20 times on each dose

SECONDARY OUTCOMES:
Plasma level of glucose | up to 2 hours after each dose
  Assessed 2 times on each dose
Plasma level of total cholesterol | up to 2 hours after each dose
  Assessed 2 times on each dose
Plasma level of C-reactive protein (CRP) | up to 2 hours after each dose
  Assessed 2 times on each dose
Plasma level of urea | up to 2 hours after each dose
  Assessed 2 times on each dose
Plasma level of creatinine | up to 2 hours after each dose
  Assessed 2 times on each dose
Plasma level of aspartate transaminase (AST) | up to 2 hours after each dose
  Assessed 2 times on each dose
Plasma level of alanine transaminase (ALT) | up to 2 hours after each dose
  Assessed 2 times on each dose
Plasma level of cortisol | up to 2 hours after each dose
  Assessed 2 times on each dose
Evaluate the subjective effects of DMT | up to 2 hours after each dose
  Assessment of the acute subjective effects of DMT by Hallucinogen Rating Scale (HRS) after each dosing. Higher scores indicate more intense psychedelic subjective effects.
Evaluate acute effects on cerebral activity using electroencephalography before, during and after the dosing | up to 2 hours after each dose
  Assessment of the electrical cerebral activity in different bandwidth as alpha, beta, theta waves by EEG before, during and after each dosing.
Assess DMT Plasma Concentration-Time Profile using High-performance liquid chromatography | up to 2 hours after each dose
  Evaluate changes in serum DMT concentration over time measured in 2, 5, 10, 15 and 120 minutes after each dosing.
Evaluate the impact of after DMT on satisfaction with life using scale | up to 1 month after dosing
  Assessment of satisfaction with life in different time points as baseline, 1, 2, 7, 14 and 28 days after dosing using the Satisfaction with Life Scale (SWL). Scores ranging from 5 to 35. Higher scores indicate greater satisfaction with life.
Evaluate the impact of DMT on trait and state of anxiety using scale | up to 1 month after dosing
  Assessment of trait and state anxiety in different time points as baseline, 1, 2, 7, 14 and 28 days after dosing using the State-Trait Anxiety Inventory (STAI). Scores ranging from 0 to 63. Higher scores indicate more severe anxiety.
Evaluate the impact of DMT on quality of life using scale | up to 1 month after dosing
  Assessment of quality of life in different time points as baseline, 14 and 28 days after dosing using the questionnaires World Health Organization Quality of Life Assessment Instrument (WHOQOL-BREF). Scores ranging from 0 to 100.
  Higher scores indicate better quality of life.
Evaluate the impact of DMT on spirituality, religiousness and personal beliefs | up to 1 month after dosing
  Assessment of spirituality, religiousness and personal beliefs in different time points as baseline, 14 and 28 days after dosing using the World Health Organization Quality of Life Assessment Instrument for Spirituality, Religiousness and Personal Beliefs (WHOQOL-SRPB). The scale is divided in 8 domains, scores ranging from 4 to 20 in each domain.
  Higher levels indicate higher level of spirituality, religiousness and personal beliefs.
Evaluate the impact of DMT on affect using scale | up to 1 month after dosing
  Assessment of affect in different time points as baseline, 1, 2, 7, 14 and 28 days after dosing using the questionnaire Positive and Negative Affect Schedule (PANAS). To score the positive affect items 1, 3, 5, 9, 10, 12, 14, 16, 17 and 19 are summed up. Scores ranging from 10 to 50. Higher scores indicate higher levels of positive affect. To score the negative affect items 2, 4, 6, 7, 8, 11, 13, 15, 18 and 20 are summed up. Scores ranging from 10 to 50. Higher scores indicate higher levels of negative affect

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário Onofre Lopes, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://biomindlabs.com